CLINICAL TRIAL: NCT04585984
Title: Effect of Antioxidant Probiotic Administration on Seminal Quality and Reproductive Outcomes.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fundación IVI (Other)
Collaborators: ADM Protexin (Industry); Biopolis S.L. (Industry); Instituto Valenciano de Infertilidad, IVI VALENCIA (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 1905-FIVI-063-NG
Record Dates: First submitted 2020-10-06; First posted 2020-10-14 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2025-08

CONDITIONS: Male Infertility
Keywords: Probiotic; Lactobacillus rhamnosus; Bifidobacterium longum; Sperm DNA fragmentation; Seminal microbiota
MeSH Terms: conditions — Infertility, Male

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The patient, investigator, assessing physician, embryologist and all site personnel with the exception of the trial nurse/coordinator and/or pharmacy assistant will remain blinded throughout the course of the trial as to which treatment each subject received.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control (Placebo Comparator): 140 men will be taking a placebo once a day during 21 days prior to the start of the IVF/ICSI cycle.
  Interventions: Dietary Supplement: Placebo
- Experimental (Experimental): 140 men will be taking the probiotic compound (50% of each probiotic: Lactobacillus rhamnosus and Bifidobacterium longum at a dose of 10^9 cfu/day) once a day for 21 days prior to the start of the IVF/ICSI cycle.
  Interventions: Dietary Supplement: Experimental - Probiotic

INTERVENTIONS:
Dietary Supplement: Experimental - Probiotic — Patients in the experimental group will take one compound (pill) a day for 21 days, containing a 50% combination of two probiotics: Lactobacillus rhamnosus and Bifidobacterium longum, at a dose of 10^9 cfu/day. The carrier of lyophilized probiotics is maltodextrin and the mixture is encapsulated in hypromellose capsules.
  Other Names: Lactobacillus rhamnosus; Bifidobacterium longum
  Arms: Experimental
Dietary Supplement: Placebo — Patients in the control group will take one unit of placebo a day for 21 days.
  Other Names: Control
  Arms: Control

SUMMARY:
The quality of semen plays a fundamental role in correct fertilization and development of normal embryos that result in a live birth. Unfortunately, semen quality has declined during the last decades, and reduced more and more. The cases of male factor infertility currently correspond to 30% of the reported cases of infertility. The parameters that are directly affected in infertile men reflecting an impaired spermatogenesis are sperm concentration, motility, morphology, ejaculate volume and DNA damage, in addition to various alterations at the molecular level that often go unnoticed and are related to the physiological capacity of the sperm. These alterations result in a decrease in reproductive capacity, which leads to the need for assisted reproduction techniques (ART). The identification of new ways to increase the quality of sperm could be very useful to improve the reproductive performance of patients.

Probiotics are defined as 'living microorganisms, which, when administered in adequate amounts, confer benefits for the health of the host'. The consumption of probiotics is increasing worldwide as therapy for many different diseases and disorders. In the field of assisted reproduction, the microbiome has been extensively studied with respect to the female endometrium to assess endometrial receptivity. However, there is little evidence about the role of the microbiome in semen. Previous studies demonstrated a moderate improvement on some sperm parameters, but still there is a need to confirm its translation into a clinical contribution to reproductive success.

The aim of this study is to evaluate the effect of these strains, Lactobacillus rhamnosus CECT8361 and Bifidobacterium longum CECT7347, on the seminal quality of infertile patients coming to IVIRMA clinics to undergo their first IVF/ICSI cycle by means of determining direct improvement on the basic sperm analysis results, on sperm DNA integrity and on the seminal microbiome profile, to ultimately evaluate the effect that it may have on the embryo quality and reproductive results of the cycles of these patients.

DETAILED DESCRIPTION:
This is a prospective randomized, unicentric, intervention study aimed at evaluating the effect of the combination of two probiotics on seminal quality and subsequent reproductive outcomes of infertile patients. As it is a food supplement, we will be subject to the Biomedicine Regulation and not to the Clinical Trials Regulation, as already classified by the Spanish Drug Agency. The study will be conducted on infertile patients at the IVIRMA Valencia clinic for two years to complete planned interventions and data collection and analysis. The reference population includes infertile patients coming to the clinic for IVF/ICSI assisted reproduction treatment with own or donated oocytes.

Patients will come to the clinic to undergo the treatment. If their characteristics are in accord with the inclusion criteria, the study will be presented and explained to them and their partners so they can evaluate their participation in it. If they wish to participate, they will sign an informed consent form, and they will be randomized using a computer-generated randomisation list into the control group (who will receive placebo) or the treatment group (who will receive the probiotic compound).

The success rate in patients with these characteristics, confirmed by the evaluation of historical information from the clinic's own database, is approximately 35% of the cycles using own oocytes, which can be used as a valid approximation. In a unilateral contrast test, assuming a risk of an alpha error of 0.05 and a beta (statistical power) of 80%, to demonstrate a difference of 15% thanks to the intervention, we need a number of 134 cases per arm and, assuming losses of 5% during the follow-up, this number would be rounded to 140 cases per study group, which makes a total of 280 couples to be included in the study.

The trial is double-blind: the patient, the investigator and all site personnel (with the exception of the trial nurse/coordinator and/or pharmacy assistant) will remain blinded throughout the course of the trial as to which treatment each subject received, including the assessing physician, the embryologist and other auxiliary members of the team.

The male assigned to the experimental group will start taking a 50% combination of the two probiotics (Lactobacillus rhamnosus CECT8361 and Bifidobacterium longum CECT7347) at a dose of 109 CFU/day on the same day of the first visit. The probiotics will be supplied by the company ADM Biopolis S.L. (Valencia, Spain). The carrier of lyophilized probiotics is maltodextrin and the mixture is encapsulated in hypromellose capsules. The patient will take one capsule daily corresponding to the administration of 109 cfu/day. The patient should take these probiotics for at least 21 days before undergoing an assisted reproduction cycle. Patients receiving the placebo will be following the same instructions. For both groups of patients, a seminal sample will be collected on their first visit to evaluate the baseline quality of the semen, as well as a microbiome analysis will be carried out using 16S rRNA sequencing (by ADM Biopolis) to determine the status of the semen at the starting point of the study. After 21 days, the patients will be appointed to deposit a second semen sample in order to perform the IVF/ICSI cycle. This sample will also be analysed, both for semen parameters and microbiome. Values obtained from both of the samples collected will be compared to observe the effect of the administration of the probiotic on the quality of sperm and its microbial population.

Fresh semen samples will be evaluated by means of a spermiogram following the standard operating procedures, in which data will be collected on volume, pH, sperm concentration, sperm mobility, cell viability and morphology. In addition, a DNA fragmentation analysis will be carried out using the Halosperm G2 kit (Halotech) based on the sperm chromatin dispersion technique. A part of the fresh sample will be frozen by submersion into liquid nitrogen and then storage in a -80ºC freezer, and sent to ADM Biopolis to perform the taxonomical identification of the bacterial populations in the semen samples using 16S rRNA sequencing with the Ion Torrent platform (Lifetechnologies).

Once the IVF/ICSI has been performed and oocytes have been correctly fertilised, embryo selection and blastocyst transfer will be carried out according to the usual medical practice to the woman's uterus, so that they can continue their development in the womb.

During recruitment, the couple will also sign a consent form allowing the team to collect data from the results of the cycle, both during embryo development and during the pregnancy and the delivery.

A database will be defined with the variables destined to be analysed according to the objectives set: semen quality analysis, sperm DNA fragmentation, microbial analysis, embryo development, gestation and delivery. The exported data will be duly codified in order to protect the clinical and personal information of the patients according to the Spanish data protection law. Finally, and prior to the statistical study, an exploratory data analysis will be carried out to review the quality of the information extracted.

The main variable of the study is the live birth rate per cycle defined as the percentage of cases in which a complete treatment of assisted reproduction is carried out with control or experimental semen, which manage to obtain offspring for each cycle of ovarian stimulation included in the study.

ELIGIBILITY:
Inclusion Criteria:

* Men aged 18-45 years old
* Men with more than 5 million progressive mobile spermatozoa in the ejaculate
* Women aged 18-37 using their own oocytes
* Women aged >37 using donated oocytes where the donor is <36 years of age.
* Women with AMH values between 1-5 ng/ml or 5-35 pmol/l

Exclusion Criteria:

* Female BMI >30kg/m^2
* Known female history of thrombophilia
* Known history of endometriosis stages III-IV
* Known history of severe adenomyosis
* Repeated implantation failures
* Recurrent miscarriages, Mullerian abnormalities or hydrosalpinx
* Use of any other probiotics by the male partner within the previous 3 months (to take account of a full spermatogenic cycle)
* Use of antibiotics by the male partner within the previous 3 months
* Known use of corticosteroids
* Known history of sexually transmitted diseases

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Semen analysis and seminal microbiota analysis.
Enrollment: 56 (Actual)
Dates: Start 2021-02-05 (Actual); Primary Completion 2024-11-14 (Actual); Study Completion 2024-11-14 (Actual)

PRIMARY OUTCOMES:
Live birth rate per cycle | through study completion, an average of 1 year
  Percentage of cases in which a complete treatment of assisted reproduction is carried out with control or experimental semen, which manage to obtain offspring for each cycle of ovarian stimulation included in the study.

CONTACTS AND LOCATIONS:
Locations (1):
- IVIRMA Valencia, Valencia, Valencia, Spain

IPD SHARING:
Plan to Share IPD: No